CLINICAL TRIAL: NCT02336490
Title: Randomized Pilot Trial of the Impact of Bedside Delivery of Discharge Medications
Brief Title: Randomized Pilot Trial of the Impact of Bedside Delivery of Discharge Medications to Pediatric Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Hatoun, General Academic Pediatric Fellow, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BostonMC
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): discharge medication prescriptions are printed or sent electronically to a patient's pharmacy of choice
- Meds-in-Hand (Active Comparator): discharge medication delivery service: discharge prescriptions are filled at the hospital pharmacy and delivered to patients before they leave the hospital
  Interventions: Other: Discharge Medication Delivery Service

INTERVENTIONS:
Other: Discharge Medication Delivery Service — hospital-owned outpatient pharmacy fills and delivers discharge medications to patients in their rooms prior to discharge
  Arms: Meds-in-Hand

SUMMARY:
This randomized pilot study proposes to field-test key logistical aspects of studying an intervention already available to patients on the pediatric ward, namely a discharge medication delivery service, called "Meds-in-Hand," which has been refined via a quality improvement process, but not rigorously studied nor fully implemented.

DETAILED DESCRIPTION:
At this time, Meds-in-Hand is not currently utilized for approximately 40% of patients admitted to the pediatric ward at Boston Medical Center. Currently patients do not receive their discharge medications via the delivery service for a variety of reasons, however they continue to receive the usual care standard employed by most hospitals, where prescriptions are sent to their home pharmacy for pickup after discharge. This study does not change the actual medications patients receive, but how and when they get them. Rigorous study of the relationship between Meds-in-Hand and patient satisfaction and clinical outcomes has not been performed to date, so there is equipoise about the value of the intervention, however observational data in the population in question, namely children admitted for an asthma exacerbation, suggest that patients who receive Meds-in-Hand prior to discharge have a reduced likelihood of a return visit to the Emergency Department in 30 days. The study will focus on parent-patient dyads admitted with an asthma exacerbation where the child is aged 2-17 years, however parents will be the exclusive study subjects. Parents of the patients will be asked a baseline, in-hospital survey as well as participate in phone follow-up interviews to report on the patient experience and parent-reported child health outcomes at approximately 3 and 30 days after leaving the hospital. 60 total parents will be enrolled, 30 in each arm of the study. This pilot study will also obtain empiric estimates of key study parameters to inform future study design and begin to examine trends between the groups of patients who are randomized to the Meds-in-Hand intervention and those randomized to usual care.

ELIGIBILITY:
Inclusion Criteria:

* admission includes treatment for asthma exacerbation
* discharge medications will require a new prescription
* primary care taker speaks english or spanish

Exclusion Criteria:

* patients being discharge outside of the operating hours of the delivery service

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Patient Experience measured by phone call followup interview | 30 days
  phone call followup interview to assess the patient experience

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hatoun, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States